CLINICAL TRIAL: NCT04904874
Title: Intense Pulsed Light Therapy in the Treatment of Refractory Meibomian Gland Dysfunction
Brief Title: Intense Pulsed Light Therapy in Meibomian Gland Dysfunction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dar Al Shifa Hospital (Other)
Responsible Party: Principal Investigator, magda torky, catract and refractie surgery specilaist, Dar Al Shifa Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02282021065726
Record Dates: First submitted 2021-05-21; First posted 2021-05-27 (Actual); Last update posted 2021-05-27 (Actual); Status verified 2021-05

CONDITIONS: Meibomian Gland Dysfunction
MeSH Terms: conditions — Meibomian Gland Dysfunction | interventions — Intense Pulsed Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- flourescein staining, miboscore (Other)
  Interventions: Device: intense pulsed light

INTERVENTIONS:
Device: intense pulsed light — treatment with 3 sessions of intense pulsed light, the second one after 2 weeks, the third one after 6 weeks

SUMMARY:
to evaluate the effect of intense pulsed light on resistant patients with Meibomian gland dysfunction

ELIGIBILITY:
Inclusion Criteria:

* age of at least 20 years.
* The diagnosis of obstructive MGD based on ocular symptoms, plugged gland oriﬁces, vascularity and irregularity of lid margins, and reduced meibum expression (meibum grade of .1, where grade 0 = clear meibum easily expressed, grade 1 = cloudy meibum expressed with mild pressure, grade 2 = cloudy meibum expressed with more than moderate pressure, and grade 3 = meibum could not be expressed even with strong pressure).
* failure of at least 3 types of conventional MGD therapy to improve symptoms or objective ﬁndings for at least 1 year before study treatment

Exclusion Criteria:

* the presence of active skin lesions, skin cancer, or other speciﬁc skin pathology.
* active ocular infection or ocular inﬂammatory disease.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Tear film break up time (TBUT) | 6 months
  After instillation of fluorescein in the conjunctival sac with fluorescein sodium strips (Jingming New TechnologicalDevelopment Co Ltd, Tianjin, China), the subject was asked to blink several times. Then, the tear film was observed under the slitlamp, using a cobalt blue filter to increase the visual contrast. For each eye, TBUT was evaluated three consecutive times, and the average of these three measurements was calculated and taken for the analysis.TBUT, a cut-off value of 5 sec was used to distinguish between moderate/severe TBUT (#5 sec) and mild/normal TBUT (.5 sec)
schirmmer staining | 6 months
  doctor places a piece of filter paper inside the lower eyelid of both eyes and the person closes their eyes.
  After 5 minutes, the doctor removes the filter paper. The doctor then assesses how far the tears have travelled on the paper. Result under 10 mm is considered to be an abnormally low level of tear production
Standard Patient Evaluation of Eye Dryness (SPEED)questionnaire | 6 months
  the self evaluated Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire (Tear Science, Morrisville, VC). This validated questionnaire asked the subject to grade the frequency and severity of four symptoms categories: (1) dryness, grittiness or scratchiness; (2) soreness or irritation; (3) burning or watering; and (4) eye fatigue. For each of these symptom categories, the subject subscored the frequency using a 4-point scale (0 never, 1 sometimes, 2 often, 3 constant), and subscored the severity using a 5-point scale (0 none, 1 tolerable, 2 uncomfortable, 3 bothersome, 4 intolerable). The SPEED score was calculated as the sum of these eight subscores. A SPEED score of 10 is widely accepted as indicating severe DED symptoms, and a cut-off value around six is often used to distinguish between asymptomatic/mild and moderate/severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Dar alshif hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No